CLINICAL TRIAL: NCT01033435
Title: The Influence of Cessation of Pomegranate Juice Intake on Inflammation and Oxidative Stress Markers and Glucose Control in Diabetic and Non Diabetic Chronic Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Dr. Ronit Geron, Deputy Head of Department, Nephrology and Hypertension Department, Western Galilee Hospital, Nahariya
Other Study IDs: Gron09
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-08

CONDITIONS: Inflammation; Oxidative Stress
Keywords: Inflammation; Oxidative stress; HbA1c; Hemodialysis
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- chronic Hemodialysis patients, treated in our unit.
  Interventions: Other: No intervention
- chronic Hemodialysis patients , No intervention: chronic Hemodialysis patients, treated in our unit.

INTERVENTIONS:
Other: No intervention
  Groups: chronic Hemodialysis patients, treated in our unit.

SUMMARY:
The current study will investigate chronic hemodialysis patients who were treated in our unit with pomegranate juice intake for 1 year - compared to a control group.

Markers will be taken 3 months after cessation of pomegranate juice intake, for inflammation and oxidative stress and Hb A1c.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Hemodialysis patients three months after termination of study which is currently carried out at our unit; which compared patients taking pomegranate juice three times a week for 1 year to a group that received placebo juice.

Exclusion Criteria:

* Patients who do not currently participate in above mentioned trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic Hemodialysis patients, treated in our unit.
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2009-12; Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Western Galilee Hospital, Nahariya, Western Galilee, Israel